CLINICAL TRIAL: NCT03355014
Title: A Randomized, Open-label, Oral Single Dosing, Two-way Crossover Clinical Trial to Compare the Safety/Tolerability and Pharmacokinetics/Pharmacodynamics of the Fixed-dose Combinations of Gemigliptin/Metformin HCl Sustained Release 50/1000 mg (25/500 mg x 2 Tablets) in Comparison to Each Component Gemigliptin 50 mg and Metformin HCl Extended Release 1000 mg (500mg x 2 Tablets) Under Fasting and Fed Conditions in Healthy Male Volunteers
Brief Title: BE Study of the Combinations of Gemigliptin/Metformin HCl Extended Release 50/1000mg(25/500mg x 2 Tablets) in Comparison to Each Component Administered Alone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LG-DMCL006
Record Dates: First submitted 2017-11-09; First posted 2017-11-28 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2017-11

CONDITIONS: Healthy Male Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemigliptin+Metformin combination therapy group (Experimental): Part I (Fasted) Combination therapy of gemigliptin/metformin sustained release 50/1000mg(25/500mg 2tablets), for 1day
  Part II (High fat diet) Combination therapy of gemigliptin/metformin sustained release 50/1000mg(25/500mg 2tablets), for 1day
  Interventions: Drug: Combination of gemigliptin/metformin HCl sustained release 50/1000mg
- Gemigliptin and Metformin coadministration therapy group (Experimental): Part I (Fasted) Coadministration therapy of gemigliptin 50mg and metformin HCL extended relese 1000mg
  Part II (High fat diet) Coadministration therapy of gemigliptin 50mg and metformin HCL extended relese 1000mg
  Interventions: Drug: Coadministration of gemigliptin 50mg and metformin HCl extended release 1000mg

INTERVENTIONS:
Drug: Combination of gemigliptin/metformin HCl sustained release 50/1000mg — Gemigliptin/Metformin HCl extended release 25/500mg 2tablets
  Arms: Gemigliptin+Metformin combination therapy group
Drug: Coadministration of gemigliptin 50mg and metformin HCl extended release 1000mg — Zemiglo 50mg 1 tablet Glucophage XR 2 tablets
  Arms: Gemigliptin and Metformin coadministration therapy group

SUMMARY:
This study is to compare the safety/tolerability and pharmacokinetics/pharmacodynamics of the fixed-dose combinations of gemigliptin/metformin HCl sustained release 50/1000 mg (25/500 mg x 2 tablets) in comparison to each component gemigliptin 50 mg and metformin HCl extended release 1000 mg (500mg x 2 tablets) under fasting and fed conditions in healthy male volunteers.

DETAILED DESCRIPTION:
This study will be conducted in separtes 2 Parts.

Part I is designed to compare the safety/tolerability and pharmacokinetics/pharmacodynamics of the fixed-dose combinations of gemigliptin/metformin HCl sustained release 50/1000 mg (25/500 mg x 2 tablets) in comparison to each component gemigliptin 50 mg and metformin HCl extended release 1000 mg (500mg x 2 tablets) under fasting condition.

Part II is designed to compare the safety/tolerability and pharmacokinetics/pharmacodynamics of the fixed-dose combinations of gemigliptin/metformin HCl sustained release 50/1000 mg (25/500 mg x 2 tablets) in comparison to each component gemigliptin 50 mg and metformin HCl extended release 1000 mg (500mg x 2 tablets) under fed conditions.

In total, 70 subjects will be enrolled in this study;Part I: 40, Part II :30 subjects.

the study design and arms are the same in both parts.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 to 45, healthy male subjects(at screening)
* Body weight between 55kg - 90kg, BMI between 18.0 - 27.0
* FPG 70-125mg/dL glucose level(at screening)
* Subjects who are appropriate to conduct study procedure in the decision of investigator
* Subject who totally understand the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress

Exclusion Criteria:

* Subject who has past or present history of any diseases following below.(liver including hepatitis virus carrier, kidney, meurology, immunology, pulmonary, endocrine, hematooncology,cardiology,mental disorder.)
* Subject who had GI tract disease or(ulcer, acute or chronic pancreatitis) surgery.(appendectomy, hernioplasty are not included)
* Subject who had drug hypersensitivity reaction.(Aspirin, antibiotics)
* Subject who already participated in other trials in 3months
* Subject who had whole blood donation in 2months, or component blood donation in 1months or transfusion in 1months currently.
* Smokers.(but, if the subject did'nt smoke in 3months, can participate the trial)

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
AUClast | up to 48hrs of post-dose(pre-dose, 0.5, 1,1.5,2,3,4,5,6,7,8,10,12,14,24,32,48, post dose at 1d and 8d)
  To evaluate AUClast of gemigliptin and metformin
Cmax | up to 48hrs of post-dose(pre-dose, 0.5, 1,1.5,2,3,4,5,6,7,8,10,12,14,24,32,48, post dose at 1d and 8d)
  To evaluate Cmax of gemigliptin and metformin

SECONDARY OUTCOMES:
AUEC | up to 48hrs of post-dose (pre-dose, 0.5, 1,1.5,2,3,4,5,6,7,8,10,12,14,24,32,48, post dose at 1d and 8d)
  This parameter is been used to measure pharmarcodynamic characters of gemigliptin and metformin, the supression rate of DPP4 activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jin X, Kim E, Huh KY, Hwang I, Cho JY, Yu KS, Lee S. Pharmacokinetics and pharmacodynamics of a fixed-dose combination of gemigliptin/metformin sustained release 25/500 mg compared to the loose combination in healthy male subjects. Transl Clin Pharmacol. 2020 Mar;28(1):43-54. doi: 10.12793/tcp.2020.28.e2. Epub 2020 Mar 30. PMID 32274380